CLINICAL TRIAL: NCT05040581
Title: Online 1-Day Cognitive Behavioural Therapy-Based Workshops for Preventing Postpartum Depression: A Pilot Study
Brief Title: 1 Day Workshops for Preventing PPD: A Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Principal Investigator, Ryan Van Lieshout, MD, PhD, Associate Professor, McMaster University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 1DayPrev
Record Dates: First submitted 2021-06-09; First posted 2021-09-10 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-02

CONDITIONS: Postpartum Depression
MeSH Terms: conditions — Depression, Postpartum

STUDY DESIGN:
Intervention Model Description: Objective 2 will be addressed using a single-group pre-post design (n=15).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Group - 1 Day CBT (Experimental): The intervention is a 6-hour long CBT-based workshop. Cognitive behavioural therapy is a structured psychotherapy based on the cognitive theory of depression that posits that negative thoughts about the self, others and the future can lead to and perpetuate depressed mood states. CBT equips participants with skills that enable them to identify and modify distortions in their thinking that lead to depressed mood and maladaptive behavioural responses.
  The intervention will be delivered in in modules and contain content on PPD etiology (with a focus on modifiable risk factors), the development of cognitive skills including cognitive restructuring, behavioural skills such as problem solving, sleep strategies, behavioural activation, assertiveness, and self-care, and the final module will involve goal setting and action planning.
  Interventions: Behavioral: 1-Day CBT-Based Workshop for Preventing PPD

INTERVENTIONS:
Behavioral: 1-Day CBT-Based Workshop for Preventing PPD — The intervention is a 6-hour long CBT-based workshop. The intervention will be delivered in in modules and contain content on PPD etiology (with a focus on modifiable risk factors), the development of cognitive skills including cognitive restructuring, behavioural skills such as problem solving, sleep strategies, behavioural activation, assertiveness, and self-care, and the final module will involve goal setting and action planning.

SUMMARY:
The aim of this pilot study is to (1) develop a treatment manual for a 1-Day CBT-Based Workshop for preventing postpartum depression that is acceptable to women; (2) recruit 15 women into a pilot workshop and seek their feedback on content, delivery and assessment procedures; and (3) conduct a small pilot randomized controlled trial (n=60) examining the impact of these workshops on rates of PPD when added to care as usual (CAU) more than CAU alone in addition to a 90-minute information session on PPD.

DETAILED DESCRIPTION:
Postpartum depression affects up to 1 in 5 mothers, however just 15% receive evidence-based treatment. It is associated with negative consequences for women and their families with enormous costs to the healthcare system. Postpartum depression is an ideal candidate for prevention because it is common, the window of opportunity to intervene is clear (pregnancy), and its risk factors are well-established and easily identifiable. Furthermore, women are in frequent contact with the healthcare system during pregnancy and are more motivated to improve their health during this time than at any other time in their lives. Given high rates of PPD and its adverse effects on mothers and their families, and the relative lack of efficient, effective psychotherapeutic interventions for preventing PPD, safe, novel, and efficient preventive interventions are needed. Since large 1-day workshops appear to successfully treat depression, given the widespread interest and investment of public health units across Canada in maternal and child health, Online 1-Day CBT-Based Workshops for Preventing PPD should be developed and tested for their ability to prevent PPD in Canadian women.

Based on longstanding clinical work with women at high risk for PPD, the development of a successful 1-Day CBT-Based Treatment Workshop for PPD and its delivery in-person and online, and an extensive review of the PPD prevention literature, the investigators will develop the content for our prevention workshop as well as an accompanying script and intervention manual for participants (Objective 1). They will then advertise and assess the feasibility of recruiting 15 women into a pilot workshop and seek their feedback on its content, delivery and assessment procedures (Objective 2). Using these data, the workshop will be revised, and the investigators will conduct a small pilot randomized controlled trial (n=60) examining the impact of these workshops on rates of PPD when added to care as usual (CAU) more than CAU alone in addition to a 90-minute information session on PPD (Objective 3).

These objectives will enable us to develop and deliver this intervention, assess the feasibility of our recruitment strategy, determine recruitment and retention rates, assess study personnel needs, refine the study protocol and estimate effect sizes for group differences in support of a larger, full-scale trial aimed as assessing the effectiveness of these workshops at reducing the likelihood of developing PPD in women at risk.

The pilot study will be considered successful and proceed to a larger trial in the future if:

1. The treatment manual for the workshop is acceptable to women
2. 15 women are recruited into a pilot workshop within three months and have 70% complete their follow-up measures
3. Recruit and randomize 60 women over six months into two separate workshop/info sessions (each consisting of 15 in the workshop and 15 into the control information session) and:

   1. 70% of eligible sign-ups enroll in the study
   2. 75% of participants assigned to experimental group complete intervention
   3. 70% of participants complete all follow-up measures
   4. Estimate a treatment effect and variance (measured using Mini International Neuropsychiatric Interview Major Depressive Disorder Module and the Edinburgh Postnatal Depression Scale)

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* >28 weeks pregnant
* do not meet diagnostic criteria for a current major depressive episode (determined using the Mini International Neuropsychiatric Interview (MINI))
* Presence of one or more of the following risk factors for PPD:
* Past history of major depressive disorder or generalized anxiety disorder (Mini International Neuropsychiatric Interview (MINI))
* Low SES (Canadian Household Low Income Cut-Off (LICOs) Before Tax)
* Single marital status (Antenatal (Psychosocial) Risk Questionnaire (ANRQ))
* Major life stress in past 12 months (Antenatal (Psychosocial) Risk Questionnaire (ANRQ))
* Major life stress in past 12 months (Antenatal (Psychosocial) Risk Questionnaire (ANRQ))
* History of physical and/or sexual abuse (Antenatal (Psychosocial) Risk Questionnaire (ANRQ))
* Perceived low social support (Antenatal (Psychosocial) Risk Questionnaire (ANRQ))

Exclusion Criteria:

* Bipolar, psychotic and/or current substance use disorders (determined using the Mini International Neuropsychiatric Interview (MINI))

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Acceptability of developed treatment manual | 6 months
  this outcome will be assessed using open-ended questions in an electronic survey to elicit participant feedback
Feasibility of recruiting 15 mothers into a pilot workshop | 6 months
  counts will be used to determine the number of participants recruited into the pilot workshop
Feasibility of recruiting 60 participants into pilot RCT in 6 months | 6 months
  counts will be used to determine the number of participants recruited into the pilot RCT
Proportion of eligible participants who enroll in study | 6 months
  counts will be used to determine the proportion of eligible participants who enroll in the study
Proportion of participants in experimental arm who complete intervention | 6 months
  counts will be used to determine the proportion of participants who complete the intervention
Proportion of participants who complete all outcome measures | 6 months
  Counts will be used to determine the number of participants who complete the outcome measures

SECONDARY OUTCOMES:
Estimate of treatment effect and variance of primary outcome for later RCT - Major Depressive Disorder | measured at 1, 2, and 3 months postpartum
  Measured using Mini International Neuropsychiatric Interview Major Depressive Disorder Module to determine if participants meet diagnostic criteria for PPD
Estimate of treatment effect and variance of primary outcome for later RCT - Depressive Symptoms | measured at 1, 2, and 3 months postpartum
  Measured using the Edinburgh Postnatal Depression Scale (EPDS) to assess level of depressive symptoms. The EPDS is a self-report measure that produces scores ranging from 0-30, with higher scores indicating higher levels of depressive symptoms. Scores of 13 or more suggest probable PPD.

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Van Lieshout, MD, PhD, Principal Investigator — McMaster University
Locations (1):
- McMaster University, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No